CLINICAL TRIAL: NCT07138573
Title: Evaluation and Comparison of the Acute Effects of Kinesio Taping Applied to the Knee and Ankle in the Lower Extremity on Balance, Proprioception, and Anterior Cruciate Ligament Injury Risk Using the Landing Error Scoring System (LESS)
Brief Title: Kinesio Taping for the Knee and Ankle: Acute Impact on Balance, Proprioception, and ACL Risk
Acronym: ACL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Zuhal Şevval Gökdere, research assistant, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2025 - 1154
Record Dates: First submitted 2025-07-23; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: ACL Injury; Kinesiotape; Balance; Proprioception; Landing Error Scoring System (LESS)
Keywords: ankle; knee; acl injury; balance; proprioception; Landing Error Scoring System (LESS); kinesiotape
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: This study is a randomized crossover trial in which each participant receives both kinesio taping interventions-one applied to the ankle and the other to the knee-with a one-week washout period between conditions. Participants are randomly assigned to either Group A (knee taping first, then ankle taping) or Group B (ankle taping first, then knee taping). Assessments are conducted immediately before and after each taping application. The study aims to compare the acute effects of taping on balance, proprioception, and ACL injury risk using standardized clinical outcome measures.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio Taping (KT) applied to the knee then ankle (Experimental): Participants receive kinesio taping on the dominant knee first, followed by ankle taping after a 1-week washout period.
  Interventions: Procedure: Kinesio Taping (KT) applied to the knee then ankle
- Kinesio Taping (KT) applied to the ankle then knee (Experimental): Participants receive kinesio taping on the dominant ankle first, followed by knee taping after a 1-week washout period.
  Interventions: Procedure: Kinesio Taping (KT) applied to the ankle then knee

INTERVENTIONS:
Procedure: Kinesio Taping (KT) applied to the knee then ankle — Procedure/Surgery: Procedure/Surgery: Kinesio Taping (KT) applied to the knee or ankle Kinesio taping was applied using a standard Y-strip with approximately 50% tension over the dominant lower extremity. In the "Knee Taping" condition, the tape was applied over the vastus medialis oblique and patellar tendon. In the "Ankle Taping" condition, the tape was applied over the peroneus longus and tibialis anterior muscles. Each taping intervention was performed by a trained physiotherapist and remained in place during the assessment session. The purpose of the intervention is to examine the acute effects of kinesio taping on balance, proprioception, and ACL injury risk using the Landing Error Scoring System (LESS).
  Arms: Kinesio Taping (KT) applied to the knee then ankle
Procedure: Kinesio Taping (KT) applied to the ankle then knee — Kinesio taping was applied using a standard Y-strip with approximately 50% tension over the dominant lower extremity. In the "Knee Taping" condition, the tape was applied over the vastus medialis oblique and patellar tendon. In the "Ankle Taping" condition, the tape was applied over the peroneus longus and tibialis anterior muscles. Each taping intervention was performed by a trained physiotherapist and remained in place during the assessment session. The purpose of the intervention is to examine the acute effects of kinesio taping on balance, proprioception, and ACL injury risk using the Landing Error Scoring System (LESS).
  Arms: Kinesio Taping (KT) applied to the ankle then knee

SUMMARY:
This study aims to evaluate and compare the acute effects of Kinesio taping applied to the knee and ankle on balance, proprioception, and anterior cruciate ligament (ACL) injury risk using the Landing Error Scoring System (LESS). Designed as a randomized crossover trial, the study will include 24 healthy volleyball athletes with at least 5 years of experience. All participants will receive both ankle and knee taping interventions, separated by a one-week washout period. Assessments will be conducted at four time points: before and after each taping. Outcome measures include the Y-Balance Test, proprioception tests, and LESS.

DETAILED DESCRIPTION:
Objective:

This study aims to evaluate and compare the acute effects of Kinesio taping applied to the knee and ankle on balance, proprioception, and anterior cruciate ligament (ACL) injury risk, assessed via the Landing Error Scoring System (LESS).

Methods:

A randomized crossover design will be used. The study will be conducted at Gazi University with 24 healthy adult volleyball athletes (≥18 years) who have been licensed players for at least 5 years. Participants will be randomly assigned to two experimental sequences:

Group A: knee taping followed by ankle taping

Group B: ankle taping followed by knee taping Each taping intervention will be separated by a one-week washout period. Assessments will be performed immediately before and after each taping session.

Knee taping will be performed using a valgus-control spiral taping technique with 50% stretch. Ankle taping will be conducted using the "figure-of-eight" method, also with 50% stretch. All applications will be administered by the same licensed physiotherapist to ensure consistency.

Outcome Measures:

Balance: Y-Balance Test (anterior, posteromedial, posterolateral reach)

Proprioception: Joint position sense tests for the knee and ankle (with eyes closed, angular replication tasks)

Injury Risk: LESS test evaluating landing biomechanics and scoring 17 specific kinematic errors

Statistical analyses will be performed using SPSS v24.0. Paired t-tests or Wilcoxon signed-rank tests will be used depending on data normality. A significance level of p<0.05 will be adopted.

Expected Results:

Kinesio taping is expected to acutely enhance proprioceptive feedback and postural control in both the knee and ankle, resulting in improved landing mechanics and a reduction in ACL injury risk. The relative effectiveness of each taping site will also be compared.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Being 18 years of age or older
* Being a licensed and regular volleyball player for at least 5 years

Exclusion Criteria:

* Being enrolled in another study or treatment program
* Being unable to complete the study for any other reason
* Having suffered a lower extremity injury within 6 months prior to participating in the study
* Female participants must be in their menstrual cycle

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Landing biomechanics score based on LESS (Landing Error Scoring System) | "Immediately after each taping intervention (same day)"
  The Landing Error Scoring System (LESS) is a reliable observational tool used to identify high-risk movement patterns associated with ACL injury. Participants will perform a standardized drop-jump task, and movement errors will be scored using the LESS protocol. A higher score indicates greater movement dysfunction and a potentially elevated risk of ACL injury. The scoring will be performed by a trained assessor using video analysis from frontal and sagittal views.

SECONDARY OUTCOMES:
Dynamic balance score based on the Y-Balance Test | "Immediately after each taping intervention (same day)"
  The Y-Balance Test is a reliable clinical tool used to assess dynamic balance and neuromuscular control of the lower extremity. Participants will be asked to perform maximal reach in three directions (anterior, posteromedial, and posterolateral) while maintaining single-leg stance on the dominant leg. The composite score will be calculated based on reach distances normalized to leg length.
Proprioception accuracy based on joint position sense | "Immediately after each taping intervention (same day)"
  Joint position sense (JPS) will be assessed using a digital inclinometer to evaluate the ability to reproduce specific knee and ankle joint angles. Participants will be blindfolded and asked to actively replicate a target angle, and the absolute angular error (in degrees) between target and replicated positions will be recorded. Lower error indicates better proprioceptive accuracy.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmapasa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to privacy concerns and institutional restrictions. The data includes sensitive health-related information, and consent for public data sharing was not obtained from participants.

REFERENCES:
- [Result] Monferrer D, Tralau T, Kertesz MA, Panjikar S, Uson I. High crystallizability under air-exclusion conditions of the full-length LysR-type transcriptional regulator TsaR from Comamonas testosteroni T-2 and data-set analysis for a MIRAS structure-solution approach. Acta Crystallogr Sect F Struct Biol Cryst Commun. 2008 Aug 1;64(Pt 8):764-9. doi: 10.1107/S1744309108019738. Epub 2008 Jul 31. PMID 18678953
- [Result] Choi SH, Lee BH, Kim HJ, Jung SW, Hwang SH, Nah SY. Differential effects of ginsenoside metabolites on slowly activating delayed rectifier K(+) and KCNQ1 K(+) channel currents. J Ginseng Res. 2013 Jul;37(3):324-31. doi: 10.5142/jgr.2013.37.324. PMID 24198658
- [Result] Treuth MS, Butte NF, Puyau M. Pregnancy-related changes in physical activity, fitness, and strength. Med Sci Sports Exerc. 2005 May;37(5):832-7. doi: 10.1249/01.mss.0000161749.38453.02. PMID 15870638
- [Result] Braith RW, Edwards DG. Exercise following heart transplantation. Sports Med. 2000 Sep;30(3):171-92. doi: 10.2165/00007256-200030030-00003. PMID 10999422
- [Result] Siparsky PN, Kocher MS. Current concepts in pediatric and adolescent arthroscopy. Arthroscopy. 2009 Dec;25(12):1453-69. doi: 10.1016/j.arthro.2009.03.011. Epub 2009 Jul 24. PMID 19962074
- [Result] Abrams PJ, Emerson CR. Rivaroxaban: a novel, oral, direct factor Xa inhibitor. Pharmacotherapy. 2009 Feb;29(2):167-81. doi: 10.1592/phco.29.2.167. PMID 19170587
- [Result] Schatz P, Moser RS, Solomon GS, Ott SD, Karpf R. Prevalence of invalid computerized baseline neurocognitive test results in high school and collegiate athletes. J Athl Train. 2012 May-Jun;47(3):289-96. doi: 10.4085/1062-6050-47.3.14. PMID 22892410
- [Result] Koitabashi K, Okamoto K, Arirto M, Sato T, Nagai K, Kurokawa MS, Suematsu N, Yasuda T, Kimura K, Kato T. Micro-sieving: isolation of whole glomeruli from a single renal needle biopsy sample. Nephron Clin Pract. 2011;117(3):c225-9. doi: 10.1159/000320198. Epub 2010 Aug 31. PMID 20805695
- [Result] Saumoy M, Jesudian AB, Aden B, Serur D, Sundararajan S, Sivananthan G, Gambarin-Gelwan M. High prevalence of colon adenomas in end-stage kidney disease patients on hemodialysis undergoing renal transplant evaluation. Clin Transplant. 2016 Mar;30(3):256-62. doi: 10.1111/ctr.12684. Epub 2016 Jan 30. PMID 26714740
- [Result] Ohji M, Okada AA, Sasaki K, Moon SC, Machewitz T, Takahashi K; ALTAIR Investigators. Correction to: Relationship between retinal fluid and visual acuity in patients with exudative age-related macular degeneration treated with intravitreal aflibercept using a treat-and-extend regimen: subgroup and post-hoc analyses from the ALTAIR study. Graefes Arch Clin Exp Ophthalmol. 2022 Jul;260(7):2395-2396. doi: 10.1007/s00417-022-05621-w. No abstract available. PMID 35366082
- [Result] Schultz H, Ying GS, Dunaief JL, Dunaief DM. Rising Plasma Beta-Carotene Is Associated With Diminishing C-Reactive Protein in Patients Consuming a Dark Green Leafy Vegetable-Rich, Low Inflammatory Foods Everyday (LIFE) Diet. Am J Lifestyle Med. 2019 Dec 21;15(6):634-643. doi: 10.1177/1559827619894954. eCollection 2021 Nov-Dec. PMID 34916884

DOCUMENTS (1):
  • Study Protocol (2025-08-13): https://cdn.clinicaltrials.gov/large-docs/73/NCT07138573/Prot_000.pdf